CLINICAL TRIAL: NCT04965467
Title: Fabry Aim Children Early (ACE) Project-Screening for Fabry Disease in a Pediatric Population at Risk
Brief Title: Fabry Aim Children Early (ACE) Project
Status: Withdrawn | Type: Observational
Why Stopped: Withdrawn due to financial reasons
Sponsor: Children's Hospital of Fudan University (Other)
Collaborators: Children's Hospital of Nanjing Medical University (Other); The Children's Hospital of Zhejiang University School of Medicine (Other); Union Hospital, Tongji Medical College, Huazhong University of Science and Technology (Other); Children's Hospital Affiliated to Zhengzhou University/Henan Children's Hospital (Unknown); Anhui Provincial Children's Hospital (Other); Beijing Children's Hospital (Other); Tianjin Children's Hospital (Other); Children's Hospital of Hebei Province (Other); Shanxi Provincial Maternity and Children's Hospital (Other); Xiamen Maternal and Child Care Hospital (Unknown); First Affiliated Hospital, Sun Yat-Sen University (Other); Children's Hospital of Chongqing Medical University (Other); West China Second University Hospital (Other); Kunming Children's Hospital (Other); Xian Children's Hospital (Other Government); Shandong Provincial Hospital (Other Government); Xinjiang Urumqi Children's Hospital. (Unknown); Hunan Children's Hospital (Other Government); Inner Mongolia Maternal and Child Healthcare Hospital (Unknown); Sichuan provincial maternity and child health care hospital (Unknown)
Responsible Party: Sponsor
Other Study IDs: ACE
Record Dates: First submitted 2021-07-08; First posted 2021-07-16 (Actual); Last update posted 2021-09-30 (Actual); Status verified 2021-09

CONDITIONS: Fabry Disease
MeSH Terms: conditions — Fabry Disease | interventions — Mass Screening

STUDY DESIGN:
Observational Model: Other | Time Perspective: Cross-Sectional
Biospecimen Retention: Samples With DNA — Whole blood
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Screening population: Screening for Fabry disease with early symptoms
  Interventions: Diagnostic Test: Screening for Fabry disease

INTERVENTIONS:
Diagnostic Test: Screening for Fabry disease — A questionnaire specifically designed to assess Fabry disease-associated phenotypes in infancy, childhood and adolescence: pain in the hands and feet, angiokeratomas, hypohidrosis, corneal whorls, unexplained renal failure, unexplained hypertrophic myocardiopathy and unexplained early onset stroke. The questionnaire consisted mainly of quantitative, closed questions with pre- defined response options.The diagnosis of FD will be performed by standard procedures following international recommendations. These require the search for a deficiency of alphagalactosidase A activity on leucocytes in males and genetic analysis of the GLA gene in females (Germain et al. 2010). In females plasma Gb3, globotriaosyl- sphingosine (lyso-Gb3) will be measured for screening.

SUMMARY:
The purpose of this study is to assess the frequency of Fabry disease in children with early symptoms.

DETAILED DESCRIPTION:
Fabry disease is a complex, multisystemic and clinically heterogeneous disease that commonly presents in childhood and is caused by deficient activity of the lysosomal enzyme alpha-galactosidaseA (α-gal A). Symptoms of Fabry disease in the pediatric population are well described. Symptoms can occur in early childhood, before age 5 years. Incidence estimations of Fabry disease vary widely. The true incidence is likely to be higher than originally thought, owing to the existence of milder variants of the disease. The purpose of this study is to assess the frequency of Fabry disease in children with early symptoms. Patients would benefit from early diagnosis, appropriate treatment, follow-up and surveillance. Early detection of Fabry patients would also benefit affected relatives, many of whom do not have a clear diagnosis of their clinical condition.

ELIGIBILITY:
Inclusion Criteria:

* Patients with fabry disease-associated phenotypes in infancy, childhood and adolescence: pain in the hands and feet, angiokeratomas, hypohidrosis, corneal whorls, unexplained renal failure, unexplained hypertrophic myocardiopathy and unexplained early onset stroke.

Exclusion Criteria:

* Patient's parent(s) or legal guardian(s) are unable to understand the nature, scope, and possible consequences of the screening.

Max Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Study Population: Patients with fabry disease-associated phenotypes in infancy, childhood and adolescence: pain in the hands and feet, angiokeratomas, hypohidrosis, corneal whorls, unexplained renal failure, unexplained hypertrophic myocardiopathy and unexplained early onset stroke.
Sampling Method: Probability Sample
Enrollment: 0 (Actual)
Dates: Start 2021-07-27 (Estimated); Primary Completion 2022-02-20 (Estimated); Study Completion 2022-02-28 (Estimated)

PRIMARY OUTCOMES:
The proportion of Fabry disease | at the enrollment
  The proportion of Fabry Disease in a defined population at risk

SECONDARY OUTCOMES:
The proportion of Fabry disease in predefined sub-populations | at the enrollment
  The proportion of Fabry Disease in a defined population at risk
The time between symptom onset and diagnosis | at the enrollment
  The time between symptom onset and diagnosis

CONTACTS AND LOCATIONS:
Locations (21):
- China (21):
  - Anhui Provincial Children's Hospital, Hefei, Anhui
  - Beijing children's hospital，capital medical university, Beijing, Beijing Municipality
  - Children's Hospital of Chongqing Medical University, Chongqing, Chongqing Municipality
  - First Affiliated Hospital, Sun Yat-Sen University, Guangzhou, Guangzhou
  - Children's Hospital of Hebei Province, Hebei, Hebei
  - Children's Hospital Affiliated to Zhengzhou University/Henan Children's Hospital, Zhengzhou, Henan
  - Wuhan Children's Hospital,Tongji Medical College, Huazhong University of Science and Technology., Wuhan, Hubei
  - Hunan Children's Hospital, Hunan, Hunan
  - Inner Mongolia Maternity and Child Healthcare Hospital, Hohhot, Inner Mongolia
  - Children's Hospital of Nanjing Medical University, Nanjing, Jiangsu
  - Kunming Children's Hospital, Kunming, Kunming
  - Shandong Provincal Hospital, Shandong, Shandong
  - Shanxi Provincial Maternity and Children's Hospital, Shanxi, Shanxi
  - West China Second University Hospital, Sichuan University, Chengdu, Sichuan
  - Sichuan provincial maternity and child health care hospital, Sichuan, Sichuan
  - Tianjin Children's Hospital, Tianjin, Tianjin Municipality
  - Xiamen Maternal and Child Care Hospital, Xiamen, Xiamen
  - Xian Children's Hospital, Xi'an, Xian
  - Xinjiang Urumqi Children's Hospital., Xinjiang, Xinjiang
  - The Children's Hospital of Zhejiang University School of Medicine, Hangzhou, Zhejiang
  - Children's Hospital of Fudan University, Shanghai

IPD SHARING:
Plan to Share IPD: Undecided